CLINICAL TRIAL: NCT00369512
Title: A Phase II Trial of Erlotinib and Radiotherapy in Patients With Stage III Cutaneous Squamous Cell Carcinomas
Brief Title: A Trial of Erlotinib + Radiotherapy for Cutaneous Squamous Cell Carcinoma
Acronym: RAD0503
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Genentech, Inc. (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Eben Rosenthal, Professor of Surgery - Otolaryngology, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F060106002
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2013-08-08 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Cancer
Keywords: Phase II; Erlotinib; Radiotherapy; Squamous Cell Carcinomas; Cutaneous; Stage III
MeSH Terms: conditions — Neoplasms; Carcinoma, Squamous Cell | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib (Experimental): Erlotinib therapy for 2 weeks (150 mg po qd)(for those who are enrolled before surgery is done), surgery/biopsy up to 8 weeks recovery, radiation/Erlotinib therapy for 6 weeks (150mg po qd).
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib therapy for 2 weeks (150 mg po qd)(for those who are enrolled before surgery is done), surgery/biopsy up to 8 weeks recovery, radiation/Erlotinib therapy for 6 weeks (150mg po qd).
  Other Names: Tarceva

SUMMARY:
This is a phase II study designed to study the effectiveness of combined radiotherapy and erlotinib in the postoperative setting for patients with cutaneous SCC that are at high risk for recurrence. Participants enrolled in the study will be evaluated by a head and neck surgeon, and a radiation oncologist. Whenever possible, a preoperative biopsy will be performed after participant enrollment in the study for histological confirmation and for molecular correlates. Participants enrolled prior to surgical resection will begin erlotinib at 150 mg by mouth (PO) every day (QD) (14 tablets) to be taken 14 days prior to surgical resection. Following planned surgical resection, the participant will begin Erlotinib therapy and radiotherapy at the same time and within 4-8 weeks of the surgical resection.

DETAILED DESCRIPTION:
This is a single-institution, open-label, non-randomized phase II trial of erlotinib administered concomitantly with radiation therapy following surgical resection of gross disease. A total of 45 patients with previously unirradiated, high-risk cutaneous SCC requiring post-operative radiotherapy will be enrolled to assess the primary endpoints of time to recurrence and disease free survival. Pretreatment biopsies will be required to confirm the histological diagnosis of SCC. Four to six weeks after surgical resection, patients will begin erlotinib (150 mg po qd) beginning the first day of radiotherapy. Patients will receive 5040 cGy beginning on day 1 of therapy in standard fractionations. Patients will be followed to evaluate for toxicity based on NCI common toxicity criteria (v3.0). Patients will be followed on protocol for a minimum of 2 years with regularly scheduled CT scans, clinical evaluations, and laboratory work. Patients with residual or recurrent cancer will be taken off protocol for salvage therapy.

As a secondary objective, molecular response of tumors to erlotinib monotherapy will be determined. When possible, participants will be enrolled and treated for 14 days with erlotinib prior to surgical resection. The pretreatment biopsy specimen (control) will then be compared to tissue acquired during the surgical resection after 14 days of erlotinib (experimental group).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven primary or recurrent squamous cell carcinoma arising from the lip or skin of the face, ear, scalp or neck.
* Participants must meet one of the four criteria:
* 1. T4 cutaneous SCC as determined by physical exam, imaging studies, prior resections or biopsy. T4 disease is defined as tumor that invades deep extradermal structures such as cartilage, skeletal muscle (e.g., muscles of facial expression), parotid gland or bone.Patients with a T2 or greater squamous cell carcinoma of the lower lip who will require post operative radiation will be allowed.
* 2. Histologically proven regional lymph node involvement (N1 disease). Fine needle aspiration or biopsy can be used to demonstrate the presence of lymphatic spread.
* 3. Histologically proven parotid gland metastasis. Fine needle aspiration or biopsy can be used to demonstrate the presence of regional spread. Includes delayed regional metastasis; primary scalp or other skin lesion treated within 36 months that would drain into the involved parotid.
* 4. Patients who following surgical resection of the primary are found to have histologically positive lymph nodes (N1). Includes delayed regional metastasis; primary lip or cutaneous lesion treated within 36 months that would drain into the involved nodal basin.
* Age > 19 years
* Tumors must be considered surgically resectable.(Patients may be enrolled after surgery is completed as long as Erlotinib therapy and concurrent radiation is started within 8 weeks of surgical resection.)
* Required laboratory data obtained prior to beginning treatment: WBC > 1,500/ml; Platelets > 90,000; serum creatinine ≤ 2.0 mg/dl
* The patient may have had a prior non-cutaneous malignancy, but must be two years from treatment.
* Performance status of ≤ 2 (ECOG scale) and life expectancy ≥ 12 months.
* The patients must agree to use effective contraception if there is the potential for procreativity. Contraception must be conducted for at least 3 months following the study.
* Patients must sign informed consent

Exclusion Criteria:

* The patient has received prior radiation therapy to the head and neck.
* The patient is pregnant or lactating
* Patients with a prior history of head and neck mucosal cancers.
* Psychological condition that renders the patient unable to understand the informed consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-08; Primary Completion 2012-01 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eben Rosenthal, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Medical Center, Birmingham, Alabama, United States

REFERENCES:
- [Result] Heath CH, Deep NL, Nabell L, Carroll WR, Desmond R, Clemons L, Spencer S, Magnuson JS, Rosenthal EL. Phase 1 study of erlotinib plus radiation therapy in patients with advanced cutaneous squamous cell carcinoma. Int J Radiat Oncol Biol Phys. 2013 Apr 1;85(5):1275-81. doi: 10.1016/j.ijrobp.2012.09.030. Epub 2012 Nov 22. PMID 23182701

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Period of recruitment was December 2006 to June 2009. Patients were screened from radiation and head/neck clinics at UAB Hospital.
Pre-assignment Details: Single Arm study
Groups:
- Erlotinib: Erlotinib therapy for 2 weeks (150 mg by mouth (PO) every day(QD))(for those who are enrolled before surgery is done), surgery/biopsy up to 8 weeks recovery, radiation/Erlotinib therapy for 6 weeks (150mg po qd).
Period: Overall Study
Arm/Group | Erlotinib
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Erlotinib: Erlotinib therapy for 2 weeks (150 mg once per day)(for those who are enrolled before surgery is done), surgery/biopsy up to 8 weeks recovery, radiation/Erlotinib therapy for 6 weeks (150mg once per day).
Arm/Group | Erlotinib
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Toxicities Associated With Combined Radiotherapy and Erlotinib Treatments.
Description: Number of gradeable toxicities (via CTCAE manual) experienced by patients on this protocol--number of events
Time Frame: 2 years
Measure: Number; unit: number of adverse events
Arm/Group | Erlotinib
Number analyzed (Participants) | 15
number of adverse events
  Dermatitis | 15
  Radiation Dermatitis | 14
  Tarceva Dermatitis | 12
  Mucositis | 13
  Esophagitis | 11
  Nausea/Vomitting | 10

2. Primary Outcome: Median Time to Cancer Recurrence
Description: Per protocol, patients were followed every 3 months for recurrent disease by physical exam and imaging (MRI/CT). Recurrence, in most cases, is detected during routine history/physical exam. If disease was detected during follow-up, every attempt was made to obtain pathological confirmation of recurrence.
Time Frame: 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 15
months | 10.5 [1 to 14]

3. Primary Outcome: Number of Patients With Recurrence at 2 Years
Description: Rate of recurrence at 2 years.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 15
participants | 4

ADVERSE EVENTS:
Time Frame: Adverse Events were reported during treatment and continued to 2 year follow-up.
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 5/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=15)
Dehydration (Metabolism and nutrition disorders) | 3
Syncope (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
CardioPulmonary Arrest (Cardiac disorders) | 1
Hematomia-Periorbital (Vascular disorders) | 1
Venous Occulsion (Vascular disorders) | 1
Cellulitis-Thigh (Musculoskeletal and connective tissue disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Weight Loss (Metabolism and nutrition disorders) | 1
Anoxeria (Metabolism and nutrition disorders) | 1
Oral Thrush (Infections and infestations) | 1
Orbital Cavity Infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib (N=15)
Dermatitis (Skin and subcutaneous tissue disorders) | 9 (15)
Oral Pain (Gastrointestinal disorders) | 2 (2)
Acneiform Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema of Flap/Lip Commissure (Skin and subcutaneous tissue disorders) | 2 (2)
Radiation Dermatitis (Skin and subcutaneous tissue disorders) | 4 (4)
Ocular/Visual (Eye disorders) | 2 (2)
Fractured Teeth (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Radiation Mucositis (Gastrointestinal disorders) | 3 (3)
Headache (Nervous system disorders) | 1 (1)
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Leg and Back Pain (General disorders) | 2 (2)
Left Chest Nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Face Pain (General disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Neuropathy CN (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No